CLINICAL TRIAL: NCT03832764
Title: Observational Study for the Evaluation of a New Non-invasive Painmonitor Used in Clinic in Awakening, Postoperative Patients
Brief Title: Non-invasive Pain Monitoring in Post-operative Patients
Acronym: ANSPEC
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/1517
Record Dates: First submitted 2018-09-11; First posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Pain, Postoperative
Keywords: skin impedance; pain monitoring; observational study; PACU/ICU
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ANSPEC-PRO: These patients are selected (after randomized selection) to be monitored non-invasively for pain level via prototype ANSPEC-PRO - correlated to a NRS number given by the awake patient in PACU/ICU.
  Interventions: Device: ANSPEC-PRO
- MEDSTORM: These patients are selected (after randomized selection) to be monitored non-invasively for pain level via MEDSTORM - correlated to a NRS number given by the awake patient in PACU/ICU.
  Interventions: Device: ANSPEC-PRO

INTERVENTIONS:
Device: ANSPEC-PRO — Device monitors for 140 minutes continuously the pain levels in awake patients in PACU/ICU
  Other Names: MEDSTORM

SUMMARY:
During the current pain monitoring system the patient is awake and he/she is asked to give a numerical scale rating from 0 (no pain) to 10 (extreme pain). The purpose is to correlate the non-invasive measurements of the prototype device ANSPEC-PRO with these numbers to develop later a method/algorithm for automatic evaluation of pain (objective measurement of pain). The measurement is done using standard ECG electrodes placed in the hand palm of the patient. The patient feels nothing during the observations, perhaps irritation of skin may occur as result of long time measurement. As a comparison to the investigators prototype, a commercial device is also used in (randomly selected) patients, i.e. the MedStorm device.

The study will try to answer the following questions:

* Are the measurements with the ANSPEC-PRO correlated with the NRS values?
* What is the (mathematical) relationship between the measured values and the NRS?
* Is there difference between the two devices in measuring pain levels? And what is this difference if pain alleviation medication is given to the patient?
* A number of 26 patients is envisaged for this study, equally distributed to be evaluated with the two devices.

ELIGIBILITY:
Inclusion Criteria:

* patients postoperative of a painfull operation
* between 18 and70 years old

Exclusion Criteria:

* day surgery patients
* chronic pain patients
* taken medication : anticonvulsants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients planned for operation, between 18 and 70 years old, not pregnant, not in chronic pain and not taken anticonvulsants or antidepressants.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Evaluation of a new non-invasive painmonitor used in clinic awakening, postoperative patients. | 140 minutes each patient
  Pain monitoring of awake patients which are standardly treated for pain using the numerical rating scale. The main outcome is a correlation between ANSPEC-PRO device and the numerical rating scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Clara Ionescu, Ghent, Oost-Vlaanderen, Belgium